CLINICAL TRIAL: NCT03360305
Title: GAPcare: The Geriatric Acute & Post-acute Care Coordination Program for Fall Prevention in the Emergency Department
Acronym: GAPcare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Elizabeth Goldberg, Assistant Professor of Emergency Medicine, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GAPcare; R03AG056349 (NIH)
Record Dates: First submitted 2017-11-27; First posted 2017-12-04 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Falls (Accidents) in Old Age
Keywords: emergency department; prevention; transitions of care
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data extractors will be blinded to the specific study arm each participant has been randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): The ED clinician will perform a standard medical evaluation. This evaluation includes a focused history and exam to identify injuries. Laboratory tests and radiologic imaging may be ordered. If necessary, the patient will receive consultation with specialty services (e.g., orthopedics). The research assistant (RA) will read the CDC STEADI brochure to the patient and provide them with a printed copy at the conclusion of their visit. The RA will solicit feedback from the clinician and the patient at the conclusion of the visit using the post-visit survey.
- Intervention (Experimental): 1. ED clinician will perform standard medical evaluation, including focused history and exam to identify injuries. RA will solicit feedback from clinician and patient via post-visit survey at conclusion of visit.
  2. PT will perform services, including integrative mobility training and lower extremity strength training and recommending outpatient services/referrals. Specific assessments and treatments will be tailored to patient.
  3. Pharmacist will perform a medication review using the updated BEERS criteria and CDC's STEADI instrument and recommend changes to potential fall risk increasing medication. Recommendations will be communicated to ED treatment team.
  4. Seniors will return home with standardized checklist containing details of their assessment and action plan. The checklist addresses patient's personal risk factors for the fall and required further actions.
  Interventions: Behavioral: GAPcare intervention

INTERVENTIONS:
Behavioral: GAPcare intervention — Subjects will receive PT and pharmacist evaluation. PT will help determine whether subject may benefit from doing exercises to improve strength or balance. PT may also supply subject with an assist device. A pharmacist will ask patient about any medication they are taking and will make recommendations on how their medication could be changed to prevent falls. Pharmacists will communicate this information to subject's doctors. Subjects will receive a fall calendar for home, where they will record any falls they have after their discharge from the ED. They will receive a phone call at home asking about any recent falls and health care interactions. Study personnel will call subjects every 2 weeks for 6 months. Subjects may receive a referral for outpatient or home-based physical and occupational therapy at the end of the visit.
  Arms: Intervention

SUMMARY:
GAPcare (Geriatric Acute & Post-acute Care Coordination Program for Fall Prevention) is an early stage investigation that enrolls older adults who present to the Emergency Department after a fall to determine the feasibility of an Emergency Department (ED)-based multidisciplinary intervention for preventing recurrent falls in older adults.

DETAILED DESCRIPTION:
Falls are the leading cause of fatal and non-fatal injury among older adults. EDs frequently evaluate older adults after their falls, but the typical evaluation consists of an injury assessment alone. There is a critical need for an ED-based intervention that addresses reasons for the fall and provides on-the-spot assessment and guidance to prevent subsequent falls. Failure to prevent subsequent falls will result in increased morbidity, mortality, healthcare utilization, loss of independence, and rising health care costs as the population of older adults increases.

Participants in GAPcare will be older adults (≥65 years-old) who present to the ED for a fall. We will pursue the following specific aims to test and further refine the GAPcare intervention: (1) Examine the feasibility of recruitment and retention of eligible patients into the GAPcare intervention, (2) determine the initial efficacy of the GAPcare intervention in reducing subsequent falls and healthcare utilization at 6 months. Our long-term goal is to prevent the early morbidity and mortality of older adults who present to the ED after a fall. The overall objective of this survey is to gather preliminary data on the feasibility of an ED based fall prevention project.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adult (non-institutionalized) 65 years-old or older presenting to ED after a fall
* Able to communicate in English
* Fall not due to syncope or external force (i.e., struck by car or assault)
* Fall not due to serious illness (i.e. stroke, acute myocardial infarction)
* Will be discharged to home, assisted living, or rehabilitation at completion of ED visit (i.e., not admitted)
* Legally authorized representative present to give informed consent if patient has cognitive impairment on Six Item Screener (score of less than four)

Exclusion Criteria:

* Unable to give informed consent due to intoxication or altered mental status
* Presence of injuries that prevent mobilization (i.e., pelvic or lower extremity fractures)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of Implementing Intervention in Emergency Department | 12 Months
  Assess the feasibility of implementing this intervention in an ED setting. We will report enrollment, reasons for accepting or declining enrollment, and drop-out from the study using the CONSORT approach. We will compare the demographic characteristics of the GAPcare participants in both arms using Chi-square or Fisher's exact test for categorical variables and Student's t-test or Wilcoxon's test for continuous variables, as appropriate. We will use Wilcoxon's test to compare the median ED length of stay between participants of both study arms.

SECONDARY OUTCOMES:
Initial efficacy | 12 Months
  Determine if the GAPcare intervention versus usual care reduces subsequent falls and all-cause and fall-related ED visits and hospital admissions in the six-month follow-up. We will compare the proportion and number of falls, ED visits, and hospital admissions in each group using chi-square (proportions) and Wilcoxon's and Student's t-tests (occurrence). If sample size permits, we will conduct survival analysis to do a time-to-event analysis. Survival time will be defined as the time from randomization to the time of the first recurrent fall, next ED visit, and hospital admission. First, we will use the Kaplan-Meier method to estimate the cumulative probability of fall-free and visit-free survival time. Next, we will use the log-rank test to test differences between survival curves for the intervention vs. usual care arm. Finally, hazard ratios and 95% confidence intervals will be calculated using the Cox Proportional Hazards model.
Feedback | 21-24 Months
  We will gather feedback from clinicians and patients on the utility and barriers of the GAPcare intervention versus usual care. We will assess 1) patient satisfaction with the care delivered, 2) barriers and facilitators of the intervention, 3) suggestions for improvement, and 4) specific feedback from clinicians on the suitability of the intervention to an ED setting. Researchers will review and code each transcript independently. A consensus process will follow, in which the researchers will categorize data into common themes within each of the 4 domains.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldberg EM, Resnik L, Marks SJ, Merchant RC. GAPcare: the Geriatric Acute and Post-acute Fall Prevention Intervention-a pilot investigation of an emergency department-based fall prevention program for community-dwelling older adults. Pilot Feasibility Stud. 2019 Aug 27;5:106. doi: 10.1186/s40814-019-0491-9. eCollection 2019. PMID 31463079
- [Result] Goldberg EM, Marks SJ, Ilegbusi A, Resnik L, Strauss DH, Merchant RC. GAPcare: The Geriatric Acute and Post-Acute Fall Prevention Intervention in the Emergency Department: Preliminary Data. J Am Geriatr Soc. 2020 Jan;68(1):198-206. doi: 10.1111/jgs.16210. Epub 2019 Oct 17. PMID 31621901
- [Derived] Goldberg EM, Marks SJ, Resnik LJ, Long S, Mellott H, Merchant RC. Can an Emergency Department-Initiated Intervention Prevent Subsequent Falls and Health Care Use in Older Adults? A Randomized Controlled Trial. Ann Emerg Med. 2020 Dec;76(6):739-750. doi: 10.1016/j.annemergmed.2020.07.025. Epub 2020 Aug 25. PMID 32854965